CLINICAL TRIAL: NCT00352053
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of Tenofovir DF as Part of an Optimized Antiretroviral Regimen in HIV-1-Infected Adolescents
Brief Title: Safety and Efficacy of Tenofovir DF in HIV-1 Infected Adolescents Failing Their Current Antiretroviral Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-104-0321
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Results first posted 2010-08-19 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-06

CONDITIONS: HIV Infections
Keywords: Phase 3; Randomized, Double-Blind; Control; Treatment-Experienced; OBR; Optimized background regimen; Highly Active Antiretroviral Therapy; HAART; HIV; HIV-1; AIDS Virus; Human Immunodeficiency Virus; Acquired Immune Deficiency Syndrome Virus; Virus; Human Immunodeficiency; Pediatrics
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Virus Diseases | interventions — Tenofovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OBR + Tenofovir DF (Experimental): Tenofovir DF administered orally, one tablet daily without regard to meals
  Interventions: Drug: Tenofovir DF
- OBR + Tenofovir DF Placebo (Placebo Comparator): Placebo to match tenofovir DF administered orally, one tablet daily without regard to meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenofovir DF — Tenofovir DF 300-mg tablet, administered orally, daily + OBR
  Arms: OBR + Tenofovir DF
Drug: Placebo — Tenofovir DF Placebo administered orally, daily + OBR
  Arms: OBR + Tenofovir DF Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of tenofovir disoproxil fumarate (tenofovir DF; TDF) plus a genotype-guided optimized background regimen (OBR) compared to placebo plus OBR in the treatment of human immunodeficiency virus type 1 (HIV-1) infected antiretroviral treatment-experienced adolescents with plasma HIV-1 ribonucleic acid (RNA) levels greater than or equal to 1000 copies/mL.

DETAILED DESCRIPTION:
This is a 48-week, randomized, double-blind, placebo-controlled, multicenter study of the safety and efficacy of tenofovir DF as part of an optimized antiretroviral regimen in HIV-1 infected adolescents (12 years to < 18 years of age) who are failing their current antiretroviral regimen and have HIV-1 RNA levels ≥ 1000 copies/mL at screening. Data from three consecutive 96-week study extensions have been used to evaluate the long-term efficacy, safety, and tolerability of open-label tenofovir DF as part of an antiviral regimen, providing data for up to 336 weeks of total drug exposure.

Pretreatment:

HIV-1 genotyping will be performed as part of the screening assessments to assist in the construction of an OBR, defined as at least 3, but no more than 5 antiretroviral agents, not including tenofovir DF or placebo.

Randomized Phase:

Participants will be randomized in a 1:1 ratio to receive either tenofovir DF + OBR, or placebo + OBR. The majority of efficacy and safety assessments will be performed at each clinic visit (Weeks 4, 8, 16, 24, 32, 40, and 48). At Week 24, participants who are adherent to study drug (in the opinion of the investigator), but do not demonstrate a ≥ 0.5 log10 copies/mL decrease from baseline in HIV-1 RNA, will be considered to be nonresponders and will be unblinded. Nonresponders randomized to the placebo group will be given the option to continue on study and receive open-label tenofovir DF with an appropriate background regimen determined by the investigator. Nonresponders randomized to the tenofovir DF treatment group will be discontinued from the study.

Extension Phases:

After completing 48 weeks of double-blind treatment with tenofovir DF or placebo, participants who have not reached 18 years of age, and who, in the opinion of the investigator, would derive clinical benefit from the use of open-label tenofovir DF, will be given the option to continue (or initiate) treatment with open-label tenofovir DF in the first of three 96 week study extension periods. Nonresponders who receive open-label tenofovir DF after Week 24 will also be considered eligible for the first study extension if they met the above criteria at Week 48.

After completing the first 96 week study extension, participants who have not reached 18 years of age, and who have shown ongoing clinical benefit from tenofovir DF, will be given the option to continue receiving open-label tenofovir DF for an additional 96 weeks or until tenofovir DF became commercially available in the country where the participants are enrolled, whichever occurs first.

After completing the second 96 week study extension, participants who have not reached 18 years of age, and who have shown ongoing clinical benefit from tenofovir DF, will be given the option to continue receiving open-label tenofovir DF for an additional 96 weeks or until tenofovir DF became commercially available in the country where the participants are enrolled, whichever occurs first.

Presentation of data:

After the randomized phase of the study, participants randomized to placebo during the randomized phase of the study and then switch to open-label tenofovir DF will have their baseline reset (defined as open-label baseline), and only outcome data collected after (on/after for adverse events (AEs)/concomitant medications) participants receive their first dose of open-label tenofovir DF will be included.

ELIGIBILITY:
Major Inclusion Criteria:

* Weight ≥ 35 kg
* Documented laboratory diagnosis of HIV infection
* Plasma HIV-1 RNA ≥ 1000 copies/mL
* Prior antiretroviral treatment experience with at least 2 antiretroviral drug classes
* Naive to tenofovir DF
* Absence of K65R mutation on genotypic testing

Exclusion Criteria:

* Patients requiring didanosine in background regimen
* Prior history of significant renal disease
* Prior history of significant bone disease

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2006-06; Primary Completion 2008-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Quirk, MD, Study Director — Gilead Sciences
Locations (18):
- Brazil (17):
  - Faculdade de Medicina - UFMG, Belo Horizonte - MG
  - Santa Casa de Belo Horizonte, Belo Horizonte - MG
  - Hospital e Maternidade Celso Pierro, Campinas - SP
  - Universidade Estadual de Campinas - UNICAMP, Campinas - SP
  - Centro de Doenças Infecciosas e Parasitárias, Campo Grande - MS
  - Hospital das Clinicas da Universidade Federal do Parana - UFPR, Curitiba - PR
  - Hospital Infantil Joana de Gusmão, Florianópolis - SC
  - Hospital Municipal Sao Jose, Joinville - SC
  - Hospital Materno Infantil Professor Fernando Figueira- IMIP, Recife
  - Hospital dos Servidores do Estado, Rio de Janeiro
  - Hospital Geral de Nova Iguacu Ambulatorio de DST e AIDS, Rio de Jeneiro
  - Hospital Guilherme Alvaro, Santos
  - Instituto da Crianca do Hospital das Clinicas da FMUSP Depto de Pediatria, Sao Paulo - SP
  - Instituto de Infectologia Emilio Ribas, Sao Paulo - SP
  - NEIMPE - Dept of Pediatrics Hospital das Clinicas FMRP-USP, São Paulo
  - Universidade Federal de Sao Paulo, Vila Clementino
  - Hospital Infantil Nossa Senhora da Gloria Servico de Infectologia Pediatria, Vitoria - ES
- Hospital del Nino, Panama City, Panama

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 17 sites in Brazil and 1 site in Panama. First participant was screened on 13 June 2006. The last study visit occurred on 19 December 2013.
Pre-assignment Details: 123 participants were screened.
Groups:
- Tenofovir DF: Tenofovir disoproxil fumarate (tenofovir DF; TDF) 300 mg tablets plus a genotype-guided optimized background regimen (OBR; 3 minimum (min.)/5 maximum (max.) antiretroviral agents (ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks.
- Placebo: Placebo to match TDF plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks.
Period: Double-Blind Phase (Through Week 48)
Arm/Group | Tenofovir DF | Placebo
Started | 45 | 42
Completed | 27 | 29 (The 10 participants discontinued for virologic failure enrolled early in the open-label extension.)
Not Completed | 18 | 13
Not completed — Virologic Failure | 14 | 10
Not completed — Physician Decision | 2 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Intolerance to Antiretroviral Regimen | 1 | 0
Period: First Extension Phase (Weeks 48-144)
Arm/Group | Tenofovir DF | Placebo
Started | 24 (3 participants completed the double-blind phase but did not enroll in the 1st extension phase.) | 36 (3 participants completed the double-blind phase but did not enroll in the 1st extension phase.)
Completed | 12 | 19
Not Completed | 12 | 17
Not completed — Physician Decision | 9 | 13
Not completed — Lack of Efficacy | 1 | 4
Not completed — Pregnancy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Second Extension Phase (Weeks 144-240)
Arm/Group | Tenofovir DF | Placebo
Started | 9 (3 participants completed the 1st extension phase but did not enroll in the 2nd extension phase.) | 14 (5 participants completed the 1st extension phase but did not enroll in the 2nd extension phase.)
Completed | 4 | 9
Not Completed | 5 | 5
Not completed — Physician Decision | 4 | 4
Not completed — Withdrawal by Subject | 1 | 1
Period: Third Extension Phase (Weeks 240-294)
Arm/Group | Tenofovir DF | Placebo
Started | 1 (3 participants completed the 2nd extension phase but did not enroll in the 3rd extension phase.) | 4 (5 participants completed the 2nd extension phase but did not enroll in the 3rd extension phase.)
Completed | 0 | 2
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study medication.
Groups:
- Tenofovir DF: TDF 300 mg tablets plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks.
- Total: Total of all reporting groups
Arm/Group | Tenofovir DF | Placebo | Total
Number analyzed (Participants) | 45 | 42 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 45 | 42 | 87
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (1.5) | 14 (1.5) | 14 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 25 | 49
  Male | 21 | 17 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 42 | 87
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 23 | 22 | 45
  Black or African Heritage | 14 | 11 | 25
  Mulatto | 4 | 4 | 8
  Mixed Race | 1 | 2 | 3
  Indian Descendant | 1 | 1 | 2
  Mestizo | 0 | 2 | 2
  Black and White Race | 1 | 0 | 1
  South American Indian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Panama | 2 | 2 | 4
  Brazil | 43 | 40 | 83
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 18.72 (2.304) | 19.99 (3.238) | 19.33 (2.849)
CD4 Cell Count [Mean (Standard Deviation); unit: cells/mm^3] | 390 (244.0) | 357 (200.8) | 374 (223.5)
CD4 Percentage [Mean (Standard Deviation); unit: Percentage of CD4 lymphocytes] — CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
  Percentage of CD4 lymphocytes | 17.8 (9.70) | 17.6 (8.31) | 17.7 (9.00)
Height [Mean (Standard Deviation); unit: cm] | 155.84 (10.071) | 156.05 (8.569) | 155.94 (9.322)
Human Immunodeficiency virus type 1 (HIV-1) ribonucleic acid (RNA) [Mean (Standard Deviation); unit: log10 copies/mL] | 4.71 (0.723) | 4.56 (0.746) | 4.64 (0.734)
Weight [Mean (Standard Deviation); unit: kg] | 45.84 (9.639) | 49.09 (11.342) | 47.41 (10.561)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Average Change From Baseline Through Week 24 (DAVG24) in Plasma HIV-1 RNA
Description: DAVG24 was defined as the time-weighted average between the first postbaseline value through the last value up to Week 24 minus the baseline value. DAVG24 was calculated using the trapezoidal rule with all available postbaseline data minus the baseline value.
  Data for participants who discontinued the randomized (double-blind) phase of the study early were included up until the point of study discontinuation (missing data not imputed).
Time Frame: Baseline to 24 Weeks
Population: Intent-to-treat (ITT) Analysis Set: participants who were randomized and received at least 1 dose of study drug, with baseline HIV-1 RNA ≥ 1000 copies/mL and who had no major eligibility criteria violations.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Groups:
- Tenofovir DF: TDF 300 mg tablets plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks. The analysis time point is calculated as the number of weeks after randomization. Only data collected during the double-blind phase are included.
- Placebo: Placebo to match TDF plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks. The analysis time point is calculated as the number of weeks after randomization. Only data collected during the double-blind phase are included.
Arm/Group | Tenofovir DF | Placebo
Number analyzed (Participants) | 44 | 41
log10 copies/mL | -1.580 [-2.15 to -0.27] | -1.549 [-2.36 to -0.34]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Time-weighted average changes from baseline through Week 24 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Time-weighted average changes from baseline through Week 24 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.55, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline genotypic sensitivity score (GSS) (without tenofovir DF) <= or > median (median GSS is 2)

2. Secondary Outcome: Time-weighted Average Change From Baseline Through Week 48 (DAVG48) in Plasma HIV-1 RNA
Description: DAVG48 was defined as the time-weighted average between the first postbaseline value through the last value up to Week 48 minus the baseline value. DAVG48 was calculated using the trapezoidal rule with all available postbaseline data minus the baseline value.
  Data for participants who discontinued the double-blind phase of the study early were included up until the point of discontinuation from the study (ie, missing data were not imputed).
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo
Number analyzed (Participants) | 44 | 41
log10 copies/mL | -1.423 [-2.25 to -0.25] | -1.352 [-2.72 to -0.53]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Time-weighted average changes from baseline through Week 48 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Time-weighted average changes from baseline through Week 48 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.40, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

3. Secondary Outcome: Change From Baseline to Week 24 in HIV-1 RNA
Time Frame: Baseline to 24 weeks
Population: ITT Analysis Set. The Tenofovir DF and Placebo groups were analyzed using the last observation carried forward (LOCF) method (includes the participant's last available postbaseline value for missing data). The Placebo/TDF groups were analyzed using the missing = excluded method (participants with missing data were excluded from the analysis).
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Groups:
- Placebo/TDF, HIV-1 RNA < 1000 Copies/mL: Participants who were randomized to placebo and switched to open-label TDF 300 mg tablets (plus OBR) with HIV-1 RNA < 1000 copies/mL at the time of the switch when a new baseline was established. The analysis time point is calculated as the number of weeks after the switch.
- Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL: Participants who were randomized to placebo and switched to open-label TDF 300 mg tablets (plus OBR) with HIV-1 RNA ≥ 1000 copies/mL at the time of the switch when a new baseline was established. The analysis time point is calculated as the number of weeks after the switch.
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 16
log10 copies/mL | -1.23 [-2.3 to -0.1] | -1.27 [-2.8 to -0.1] | 0.0 [0.0 to 0.0] | -0.1 [-0.6 to 0.3]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 24 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 24 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.58, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

4. Secondary Outcome: Change From Baseline to Week 48 in HIV-1 RNA
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set. The Tenofovir DF and Placebo groups were analyzed using the LOCF method. The Placebo/TDF groups were analyzed using the missing = excluded method.
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 8
log10 copies/mL | -0.97 [-2.3 to 0.0] | -1.53 [-3.0 to 0.0] | 0.0 [0.0 to 0.6] | 0.2 [-0.1 to 0.5]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 48 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 48 in plasma HIV-1 RNA for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.37, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

5. Secondary Outcome: Change From Baseline to Week 96 in HIV-1 RNA
Time Frame: Baseline to 96 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Groups:
- Tenofovir DF: TDF 300 mg tablets plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks. The analysis time point is calculated as the number of weeks after randomization.
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 19 | 17 | 3
log10 copies/mL | -2.1 [-2.5 to -0.6] | 0.0 [0.0 to 0.9] | 0.1 [-1.4 to 0.8]

6. Secondary Outcome: Change From Baseline to Week 144 in HIV-1 RNA
Time Frame: Baseline to 144 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 10 | 11 | 2
log10 copies/mL | -2.5 [-2.7 to -2.2] | 0.2 [0.0 to 1.6] | 0.7 [0.6 to 0.8]

7. Secondary Outcome: Change From Baseline to Week 192 in HIV-1 RNA
Time Frame: Baseline to 192 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 5 | 2
log10 copies/mL | -2.0 [-2.5 to -0.7] | 0.0 [0.0 to 0.2] | -0.1 [-1.4 to 1.3]

8. Secondary Outcome: Change From Baseline to Week 240 in HIV-1 RNA
Time Frame: Baseline to 240 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 4 | 2 | 1
log10 copies/mL | -2.5 [-2.6 to -2.2] | -0.4 [-0.8 to 0.0] | -1.4 [-1.4 to -1.4]

9. Secondary Outcome: Change From Baseline to Week 288 in HIV-1 RNA
Time Frame: Baseline to 288 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: log10 copies/mL
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
log10 copies/mL | -1.1 [-1.1 to -1.1] | -0.8 [-0.8 to -0.8] | 0.6 [0.6 to 0.6]

10. Secondary Outcome: Change From Baseline to Week 336 in HIV-1 RNA
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Baseline to 336 weeks
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline to Week 24 in Cluster Determinant 4 (CD4) Count
Time Frame: Baseline to 24 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 42 | 41 | 18 | 16
cells/mm3 | 69 [-26 to 172] | 49 [-3 to 156] | -43 [-181 to 53] | -12 [-48 to 59]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 24 in plasma CD4 count for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 24 in CD4 count for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.71, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

12. Secondary Outcome: Change From Baseline to Week 48 in CD4 Count
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 32 | 31 | 17 | 11
cells/mm3 | 152 [-4 to 241] | 148 [42 to 289] | 15 [-69 to 95] | -47 [-83 to 67]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 48 in plasma CD4 count for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 48 in CD4 count for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.47, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

13. Secondary Outcome: Change From Baseline to Week 96 in CD4 Count
Time Frame: Baseline to 96 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 20 | 17 | 3
cells/mm3 | 152 [52 to 266] | -6 [-96 to 85] | -69 [-75 to 278]

14. Secondary Outcome: Change From Baseline to Week 144 in CD4 Count
Time Frame: Baseline to 144 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 12 | 11 | 2
cells/mm^3 | 188 [53 to 361] | -88 [-165 to 93] | 33 [-109 to 174]

15. Secondary Outcome: Change From Baseline to Week 192 in CD4 Count
Time Frame: Baseline to 192 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 6 | 2
cells/mm^3 | 166 [-82 to 333] | -70 [-155 to 220] | -23 [-46 to 1]

16. Secondary Outcome: Change From Baseline to Week 240 in CD4 Count
Time Frame: Baseline to 240 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 5 | 2 | 1
cells/mm^3 | 221 [59 to 368] | 571 [-13 to 1155] | 258 [258 to 258]

17. Secondary Outcome: Change From Baseline to Week 288 in CD4 Count
Time Frame: Baseline to 288 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
cells/mm^3 | 310 [310 to 310] | 100 [100 to 100] | 309 [309 to 309]

18. Secondary Outcome: Change From Baseline to Week 336 in CD4 Count
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Baseline to 336 weeks
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Change From Baseline to Week 24 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 24 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 42 | 41 | 18 | 16
Percentage of CD4 lymphocytes | 3.0 [0.0 to 6.0] | 2.0 [-1.0 to 4.0] | 0.0 [-3.0 to 3.0] | -1.0 [-3.0 to 2.0]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 24 in plasma CD4% for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 24 in CD4% for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.26, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

20. Secondary Outcome: Change From Baseline to Week 48 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 48 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 32 | 31 | 17 | 11
Percentage of CD4 lymphocytes | 6.0 [2.5 to 9.0] | 5.0 [2.0 to 8.0] | 2.0 [1.0 to 4.0] | -1.0 [-4.0 to 7.0]
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Changes from baseline through Week 48 in plasma CD4% for the tenofovir DF and placebo groups are equal. Alternative hypothesis: Changes from baseline through Week 48 in CD4% for the tenofovir DF and placebo groups are different (two-sided); Test type: Superiority or Other; p = 0.63, Van Elteren test — No adjustments for multiple comparisons were made; P-value is from a Van Elteren test stratified by baseline GSS (without tenofovir DF) <= or > median (median GSS is 2)

21. Secondary Outcome: Change From Baseline to Week 96 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 96 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 20 | 17 | 3
Percentage of CD4 lymphocytes | 5.0 [2.0 to 8.0] | 2.0 [0.0 to 5.0] | 9.0 [2.0 to 15.0]

22. Secondary Outcome: Change From Baseline to Week 144 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 144 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 12 | 11 | 2
Percentage of CD4 lymphocytes | 6.5 [-2.0 to 13.0] | 0.0 [-4.0 to 8.0] | 5.5 [2.0 to 9.0]

23. Secondary Outcome: Change From Baseline to Week 192 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 192 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 6 | 2
Percentage of CD4 lymphocytes | 5.0 [-2.0 to 11.6] | 1.9 [-1.0 to 10.0] | 4.8 [1.5 to 8.0]

24. Secondary Outcome: Change From Baseline to Week 240 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 240 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 5 | 2 | 1
Percentage of CD4 lymphocytes | 10.0 [-2.0 to 13.3] | 8.9 [8.2 to 9.6] | 18.9 [18.9 to 18.9]

25. Secondary Outcome: Change From Baseline to Week 288 in CD4 Percentage
Description: CD4 percentage is the percentage of total lymphocytes that are CD4 cells.
Time Frame: Baseline to 288 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Median (Inter-Quartile Range); unit: Percentage of CD4 lymphocytes
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
Percentage of CD4 lymphocytes | 7.4 [7.4 to 7.4] | 4.0 [4.0 to 4.0] | 11.9 [11.9 to 11.9]

26. Secondary Outcome: Change From Baseline to Week 336 in CD4 Percentage
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Baseline to 336 weeks
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 24
Time Frame: Baseline to 24 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 16
Percentage of participants | 56.8 | 51.2 | 0 | 12.5
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants who had at least a 1.0 log10 copies/mL decrease from baseline to Week 24 in HIV-1 RNA for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants who had at least a 1.0 log10 copies/mL decrease from baseline to Week 24 in HIV-1 RNA for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 0.67, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

28. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 48
Time Frame: Baseline to 48 weeks
Population: as for outcome 4
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 8
Percentage of participants | 47.7 | 53.7 | 0 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants who had at least a 1.0 log10 copies/mL decrease from baseline to Week 48 in HIV-1 RNA for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants who had at least a 1.0 log10 copies/mL decrease from baseline to Week 48 in HIV-1 RNA for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 0.67, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

29. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 96
Time Frame: Baseline to 96 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 19 | 17 | 3
Percentage of participants | 73.7 | 5.9 | 33.3

30. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 144
Time Frame: Baseline to 144 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 10 | 11 | 2
Percentage of participants | 90.0 | 0 | 0

31. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 192
Time Frame: Baseline to 192 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 5 | 2
Percentage of participants | 71.4 | 0 | 50.0

32. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 240
Time Frame: Baseline to 240 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 4 | 2 | 1
Percentage of participants | 100.0 | 0 | 100.0

33. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0log 10 Copies/mL From Baseline to Week 288
Time Frame: Baseline to 288 weeks
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
Percentage of participants | 100.0 | 0 | 0

34. Secondary Outcome: Percentage of Participants With an HIV-1 RNA Decrease of ≥ 1.0 log10 Copies/mL From Baseline to Week 336
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Baseline to 336 weeks
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 24
Time Frame: Week 24
Population: ITT Analysis Set. The Tenofovir DF and Placebo groups were analyzed using the missing = failure method in which participants with missing data were considered to have failed to achieve the endpoint. The Placebo/TDF groups were analyzed using the missing = excluded method.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 16
Percentage of participants | 40.9 | 41.5 | 83.3 | 6.3
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 24 for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 24 for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 1.00, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

36. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 48
Time Frame: Week 48
Population: ITT Analysis Set. The Tenofovir DF and Placebo groups were analyzed using the missing = failure method. The Placebo/TDF groups were analyzed using the missing = excluded method.
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 8
Percentage of participants | 34.1 | 43.9 | 77.8 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants with HIV-1 RNA < 400 copies/mL at Week 48 for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 0.38, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

37. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 96
Time Frame: Week 96
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 19 | 17 | 3
Percentage of participants | 63.2 | 70.6 | 33.3

38. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 144
Time Frame: Week 144
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Groups:
- Placebo/TDF, HIV-1 RNA >= 1000 Copies/mL: Participants who were randomized to placebo and switched to open-label TDF 300 mg tablets (plus OBR) with HIV-1 RNA ≥ 1000 copies/mL at the time of the switch when a new baseline was established. The analysis time point is calculated as the number of weeks after the switch.
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA >= 1000 Copies/mL
Number analyzed (Participants) | 10 | 11 | 2
Percentage of participants | 70.0 | 72.7 | 0

39. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 192
Time Frame: Week 192
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 5 | 2
Percentage of participants | 57.1 | 80.0 | 50.0

40. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 240
Time Frame: Week 240
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 4 | 2 | 1
Percentage of participants | 75.0 | 100.0 | 100.0

41. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 288
Time Frame: Week 288
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
Percentage of participants | 0 | 100.0 | 0

42. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 400 Copies/mL at Week 336
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Week 336
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

43. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24
Time Frame: Week 24
Population: as for outcome 36
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 16
Percentage of participants | 20.5 | 34.1 | 77.8 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 0.22, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

44. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48
Time Frame: Week 48
Population: as for outcome 36
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 44 | 41 | 18 | 8
Percentage of participants | 27.3 | 36.6 | 61.1 | 0
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 for the tenofovir DF and placebo groups is equal. Alternative hypothesis: Percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 for the tenofovir DF and placebo groups is different (two-sided); Test type: Superiority or Other; p = 0.48, Fisher Exact — No adjustments for multiple comparisons were made; No adjustments were made

45. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96
Time Frame: Week 96
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 19 | 17 | 3
Percentage of participants | 47.4 | 58.8 | 33.3

46. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 144
Time Frame: Week 144
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 10 | 11 | 2
Percentage of participants | 70.0 | 45.5 | 0

47. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 192
Time Frame: Week 192
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 7 | 5 | 2
Percentage of participants | 42.9 | 60.0 | 50.0

48. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 240
Time Frame: Week 240
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 4 | 2 | 1
Percentage of participants | 75.0 | 100.0 | 100.0

49. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 288
Time Frame: Week 288
Population: ITT Analysis Set, missing = excluded method
Measure: Number; unit: Percentage of participants
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 1 | 1 | 1
Percentage of participants | 0 | 100.0 | 0

50. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 336
Description: No analysis was performed because the last study participant discontinued after Week 294 and the study was closed.
Time Frame: Week 336
Population: ITT Analysis Set, missing = excluded method
Arm/Group | Tenofovir DF | Placebo/TDF, HIV-1 RNA < 1000 Copies/mL | Placebo/TDF, HIV-1 RNA ≥ 1000 Copies/mL
Number analyzed (Participants) | 0 | 0 | 0

51. Secondary Outcome: Percentage of Participants With Virologic Failure Through Week 48
Description: Virologic failure was defined as either nonresponse or viral rebound.
  * Nonresponse (failure to achieve response). Response was defined as either
    * A ≥ 0.5 log10 copies/mL decrease in HIV-1 RNA from baseline at 2 consecutive visits, or
    * HIV-1 RNA < 400 copies/mL at 2 consecutive visits.
  * Viral rebound was defined as either
    * Participants who achieved a ≥ 0.5 log10 copies/mL decrease from baseline in plasma HIV-1 RNA at 2 consecutive visits, who then subsequently achieved plasma HIV-1 RNA values ≥ 1.0 log10 copies/mL above their on-study nadir (lowest value) and/or plasma HIV-1 RNA values ≥ the baseline value at 2 consecutive visits, or
    * Participants who achieved plasma HIV-1 RNA levels of < 400 copies/mL at 2 consecutive visits, and then subsequently had plasma HIV-1 RNA levels > 1000 copies/mL at 2 consecutive visits.
  The virologic failure rate was estimated from Kaplan-Meier product limit method by including all HIV-1 RNA data collected during the double-blind phase.
Time Frame: Up to 48 weeks
Population: ITT Analysis Set. 1 participant without time to respond [6 days of treatment]) was excluded. Nonresponders were counted as failures at time 0. Rebounders were counted as failures on study day of the first of 2 assessments meeting criteria. Otherwise, they were censored at last double-blind HIV measurement.
Measure: Number; unit: Kaplan-Meier percentage
Groups:
- Placebo: Placebo to match TDF plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks. The analysis time point is calculated as the number of weeks after randomization.
Arm/Group | Tenofovir DF | Placebo
Number analyzed (Participants) | 43 | 41
Kaplan-Meier percentage | 51 | 39
Statistical Analysis 1: Comparison: Tenofovir DF vs Placebo; Null hypothesis: The survival functions for the tenofovir DF and placebo groups up to Week 48 are equal. Alternative hypothesis: The survival functions for the tenofovir DF and placebo groups up to Week 48 are different (two-sided); Test type: Superiority or Other; p = 0.29, Log Rank — No adjustments for multiple comparisons were made; No adjustments were made

ADVERSE EVENTS:
Time Frame: Up to Week 294 plus 30 days.
Description: Safety Analysis Set: participants were randomized and received at least 1 dose of study medication. MedDRA version 11.1 was used for the Tenofovir DF and Placebo columns; MedDRA version 16.1 was used for the All TDF column.
Groups:
- Tenofovir DF: Adverse events occurring in the double-blind phase are presented for this reporting group.
  TDF 300 mg tablets plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks.
- Placebo: Adverse events occurring in the double-blind phase are presented for this reporting group.
  Placebo to match TDF plus a genotype-guided OBR (3 min./5 max. ARVs) from baseline to Week 48 (double-blind phase), followed by open-label TDF 300 mg plus OBR for up to an additional 288 weeks.
- All TDF: Adverse events reported for the All TDF group include those reported during the double-blind phase and/or extension phase for subjects who were randomized to TDF group plus adverse events reported during the extension phase only for subjects who switched from placebo to open-label TDF.
  Tenofovir DF 300-mg tablets in participants initially randomized to the Tenofovir DF group, and in those initially randomized to the Placebo group who later switched to open-label TDF 300 mg.
Arm/Group | Tenofovir DF | Placebo | All TDF
Serious Adverse Events (participants affected / at risk) | 10/45 | 3/42 | 20/81
Other Adverse Events (participants affected / at risk) | 44/45 | 35/42 | 76/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=45) | Placebo (N=42) | All TDF (N=81)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 5
Sinusitis (Infections and infestations) | 2 | 0 | 2
Herpes Zoster (Infections and infestations) | 0 | 0 | 3
Cryptococcosis (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1
Pneumocystis Jiroveci Pneumonia (Infections and infestations) | 2 | 0 | 2
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1
Abscess Limb (Infections and infestations) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cerebral Toxoplasmosis (Infections and infestations) | 0 | 1 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Neurocryptococcosis (Infections and infestations) | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 0 | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tenofovir DF (N=45) | Placebo (N=42) | All TDF (N=81)
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 7
Conjunctivitis (Eye disorders) | 2 | 1 | 5
Vomiting (Gastrointestinal disorders) | 16 | 5 | 21
Diarrhoea (Gastrointestinal disorders) | 10 | 4 | 17
Nausea (Gastrointestinal disorders) | 11 | 3 | 15
Abdominal Pain (Gastrointestinal disorders) | 8 | 5 | 9
Gastritis (Gastrointestinal disorders) | 5 | 1 | 7
Constipation (Gastrointestinal disorders) | 3 | 0 | 4
Pyrexia (General disorders) | 4 | 5 | 7
Jaundice (Hepatobiliary disorders) | 3 | 3 | 4
Sinusitis (Infections and infestations) | 12 | 6 | 24
Nasopharyngitis (Infections and infestations) | 8 | 7 | 18
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 3 | 17
Tonsillitis (Infections and infestations) | 4 | 3 | 12
Oral Herpes (Infections and infestations) | 5 | 3 | 9
Tracheobronchitis (Infections and infestations) | 5 | 1 | 9
Acute Sinusitis (Infections and infestations) | 3 | 4 | 6
Rhinitis (Infections and infestations) | 3 | 1 | 7
Pneumonia (Infections and infestations) | 2 | 2 | 5
Body Tinea (Infections and infestations) | 2 | 1 | 5
Furuncle (Infections and infestations) | 3 | 1 | 4
Gastroenteritis (Infections and infestations) | 2 | 1 | 5
Bronchopneumonia (Infections and infestations) | 2 | 0 | 5
Hordeolum (Infections and infestations) | 3 | 1 | 3
Impetigo (Infections and infestations) | 1 | 3 | 3
Herpes Zoster (Infections and infestations) | 0 | 3 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 3 | 6
Anorexia (Metabolism and nutrition disorders) | 4 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 5
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 5
Skin Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 2
Headache (Nervous system disorders) | 6 | 5 | 16
Dizziness (Nervous system disorders) | 8 | 5 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 24
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 7

LIMITATIONS AND CAVEATS:
Participants left the study for a number of reasons (eg, turned 18 years old, switched to a different HIV treatment regimen), which led to small numbers of participants analyzed at later time points, and the study was concluded earlier than planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years